CLINICAL TRIAL: NCT00657722
Title: Identification Of The Predictive Angiographic And Computed Tomographic (CT) Criteria Of The Success Of The Thromboendarterectomy In Chronic Pulmonary Hypertension
Brief Title: Identification of Criteria of the Success of the Endarterectomy in Chronic Pulmonary Post Embolic Hypertension
Acronym: ETHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: K060205
Record Dates: First submitted 2008-03-28; First posted 2008-04-14 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Pulmonary hypertension; Chronic thromboembolic pulmonary hypertension; Operability; Thromboendarteriectomy; Operative mortality rate; Technical failure; Pulmonary angiography; Computed tomography
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — homeobox protein PITX3

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Angiography and Computed Tomography
  Interventions: Other: Angiography and Computed Tomography

INTERVENTIONS:
Other: Angiography and Computed Tomography — Preoperative angiography and Computed Tomography
  Other Names: standardized reading grids of APN and ASMD

SUMMARY:
In order to improve effectiveness of the surgical operation thanks to a reduction in the rate of failure, this study will allow us to identify predictive angiographic and CT finding of surgical failure, starting from standardized reading grids, in order to have a better selection of the operable patients.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension(CTEPH) is caused by obstruction of the large pulmonary arteries by acute and recurrent pulmonary emboli, and organization of these blood clots. ANTOINE BECLERE respiratory unit, in partnership with the MARIE LANNELONGUE hospital thoracic and vascular surgery departments was designated recently as reference national centre for pulmonary hypertension and represents the only French structure for evaluation of CTEPH with 150 patients addressed each year.If the disease is proximately located, CTEPH can be cured surgically through a complex surgical procedure performed under Hypothermia and total circulatory arrest. In spite of multidisciplinary meeting deciding the operability of each case the rate of failure is approximately of 15% (9% of operative mortality rate and 6% of technical failure).

The aim of this study is to identify predictive angiographic and CT findings of success, by allowing a better selection of operable patients.

It would be possible to improve the effectiveness of the surgical treatment and reduce the rate failure from 15% to 7 % or even 5 %.

ELIGIBILITY:
Inclusion Criteria:

* Patients addressed to the reference centre of pulmonary hypertension for a suspected CPC-PE
* Achieving an assessment prior to the operation, including:1) Right cardiac catheterization confirming HTP with a mean pulmonary arterial pressure> 25 mm Hg at rest; 2) Echography and Doppler of the lower limbs in search of phlebitis sequela; 3) Pulmonary scintigraphy with 6 views in ventilation and perfusion; 4) Digital pulmonary angiography; 5) A 64 detector pulmonary computed tomography; 6) Having read the briefing note and given their agreement.

Exclusion criteria:

* Refusal examinations .
* Patient for which one method is contraindicated
* Patient considered not operable by the staff
* Life expectancy of less than 3 months
* Geographical distance for the clinical follow-up at 3 months
* Renal insufficiency (creatinine clearance <30 mL / min)
* Proven allergy to iodinated contrast agents
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2008-01; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
surgical effectiveness evaluated by the death or failure rate. | 6 months

SECONDARY OUTCOMES:
surgical effectiveness evaluated by the death or failure rate. | 3 months
Check that none of the patients considered unresectable on data from staff was declared operable with the criteria predictive success of imaging examinations. | before surgery
Determine the interest of pulmonary angiography in the operability decision compared first to Multi detector AngioCT alone with standardized analyze and then with the both exams. | before surgery
Determine the incidence of adverse events associated with each of these two exams or their combination. | 3 and 6 months after surgery
Check-inter-observer reproducibility of standardized reading grids of pulmonary angiography and MD-AngioCT | Before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu LIBERATORE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère; Dominique MUSSET, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris, Hôpital Antoine Béclère; Gerald SIMONNEAU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris, Hôpital Antoine Béclère
Locations (2):
- France (2):
  - Hôpital Antoine Beclere, Clamart
  - Hospital Marie Lannelongue, Le Plessis-Robinson